CLINICAL TRIAL: NCT06347146
Title: Bridges2Scale: Testing Implementation Strategies for an Economic Empowerment Intervention Among Young People Orphaned by AIDS
Brief Title: Bridges2Scale: Testing Implementation Strategies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD112323 (NIH); R01HD112323 (NIH)
Record Dates: First submitted 2024-03-17; First posted 2024-04-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard implementation strategy condition (Experimental): The Standard Implementation strategy condition is one that has been applied in our prior randomized controlled trials (RCTs). In applying this strategy, the investigators will meet with both non-governmental organizations (NGO) and school staff to gauge NGOs interest in partnering on study implementation and describe roles and responsibilities.
  Interventions: Behavioral: Financial Literacy Training (FLT) workshops; Behavioral: Mentorship; Behavioral: Income Generation Activity (IGA); Behavioral: Youth Development Accounts (YDA)
- Enhanced Implementation strategy condition (Experimental): The Enhanced Implementation strategy condition will be developed using Implementation Mapping, a systematic protocol for developing implementation strategies using theory, evidence, and stakeholder input. This will ensure that known determinants of implementation, scale-up, and sustainment are addressed by strategies designed collaboratively with the community partners from a public-private partnership of government-funded public schools and non-government organizations (NGOs).
  Interventions: Behavioral: Financial Literacy Training (FLT) workshops; Behavioral: Mentorship; Behavioral: Income Generation Activity (IGA); Behavioral: Youth Development Accounts (YDA)

INTERVENTIONS:
Behavioral: Financial Literacy Training (FLT) workshops — Adolescents and youths and their caregivers will receive six 1-2 hour workshop sessions that cover components on saving, and financial management. The sessions will: introduce participants to saving, saving strategies, career planning, and the utilization of financial institutions, including saving in banks.
  Other Names: FLT workshops
Behavioral: Mentorship — Each adolescent and youth will have a mentor who will visit with them monthly for the duration of the intervention. The one-to-one mentorship program is intended to help AYaAIDS overcome a variety of challenges they face in daily life by fostering meaningful and lasting relationships with near peer or adult role models. Resilience theory posits that having a supportive adult outside the family reduces the impact of stress on AY's mental health. Mentors will be high school students who will be trained by the schools or NGO staff depending on study condition. All mentors will be reimbursed for their transport expenses to the field, plus an equivalent of a $5 gift card for airtime per visit.
Behavioral: Income Generation Activity (IGA) — Participants will be trained on investing in income-generating activities (IGA) during the FLT workshops and will be allowed to use up to 30% of their matched savings to invest in an IGA intended to benefit the adolescent and youth (AY) and their caregiving families. The IGA portion is intended to promote economic stability.
Behavioral: Youth Development Accounts (YDA) — Each adolescent and youth (AY) will receive a youth development account, which is a matched savings account held in the AY's name in a financial institution under the Central Bank (Bank of Uganda). Any of the AY's family members, relatives, or friends is encouraged to contribute towards the YDA. The account is then matched with money from the program. The match cap (maximum family contribution to be matched by the program) will be an equivalent of US$10 a month per family or US$200 for the 20-months intervention period. AY who save the maximum amount will have $600 ($200 plus $400 in match-a 2:1 match rate).

SUMMARY:
The goal of this clinical trial is to compare two multifaceted strategies (standard vs enhanced) for scaling Bridges in a two-arm Hybrid III effectiveness-implementation cluster randomized controlled trial (RCT) in adolescent and youths affected by AIDS [AYaAIDS] (ages 11-17 years) from 48 schools in the Greater Masaka region of Uganda. The main aims of the clinical trial are: Aim 1. Compare the implementation effectiveness of the standard implementation strategy vs. an enhanced implementation strategy. The investigators will assess fidelity to Bridges (primary implementation outcome) and sustainment of Bridges (exploratory implementation outcome).

Aim 2. Determine the clinical effectiveness of Bridges implemented via a standard vs. enhanced implementation strategy. Aim 3: Explore implementation processes, mechanisms, and determinants. Aim 4. Compare the cost and cost-effectiveness of the two implementation strategies. Using an activity-based ingredients approach, the investigators will examine how much each strategy costs to achieve a unit of effect.

DETAILED DESCRIPTION:
Economic empowerment (EE) interventions have demonstrated substantial promise in reducing HIV-related risk-taking behaviors, and improving ART treatment adherence and mental health outcomes. Our group has demonstrated the effectiveness of a multi-component EE intervention, Bridges, in four NIH-funded randomized control trials (RCT) in Uganda. Bridges involves: 1) financial literacy training (FLT) and mentorship; 2) family income-generating activities (IGA); and 3) incentivized savings via a matched Youth Development Account (YDA) for education, family small business investment, and/or health-related expenses. Bridges has demonstrated robust effects on HIV-related risk-taking behaviors, antiretroviral therapy (ART) adherence, mental health, psychosocial outcomes, educational achievement, family economics, and family cohesion. Yet, scaling EE interventions has been a challenge, signaling the need to identify and test implementation strategies and examine determinants of implementation and sustainment. In Bridges2Scale, the goal of this clinical trial is to compare two multifaceted strategies (standard vs enhanced) for scaling Bridges in a two-arm Hybrid III effectiveness-implementation cluster RCT in adolescent and youths affected by AIDS [AYaAIDS] (ages 11-17 years) from 48 schools in the Greater Masaka region of Uganda. The main aims of the clinical trial are:

Aim 1. Compare the implementation effectiveness of the standard implementation strategy vs. an enhanced implementation strategy. The investigators will assess fidelity to Bridges (primary implementation outcome) and sustainment of Bridges (exploratory implementation outcome).

Aim 2: Determine the clinical effectiveness of Bridges implemented via a standard vs. enhanced implementation strategy. The investigators will assess HIV prevalence (primary outcome measured via participants' HIV status). In exploratory analyses, the investigators will assess economic stability, school attendance and attainment, sexual risk-taking behavior, mental health functioning, viral suppression (for AYLHIV), and pre-exposure prophylaxis (PrEP) use (for HIV-negative adolescents). Participants from each of the 48 schools will be randomly assigned to one of the two study conditions (n=720 participants; n=24 schools per study condition) such that all selected children from a particular school will receive the same intervention to reduce contamination. After the baseline assessment, data will be collected at 4 follow-up time points (12 months, 24 months, 36 months, and 48 months). The investigators will compare the implementation effectiveness (mean levels of fidelity) of the standard implementation strategy to the enhanced strategy and compare whether adolescents in the enhanced implementation strategy will have a lower odds of HIV prevalence at the final measurement point (48 months). The investigators will also compare the superiority of the enhanced implementation strategy to the standard implementation strategy group in lowering sexual risk-taking behavior, improving economic stability, education related outcomes (school attendance and attainment), and mental health functioning (for all adolescents), viral suppression (for AYLHIV), and PrEP use (for HIV negative adolescents).

Aim 3: Explore implementation processes, mechanisms, and determinants. Using mixed methods, the investigators will apply standardized measures and semi-structured interviews with implementing teams to explore any modifications to the two implementation strategies, perceptions of the implementation strategies (acceptability, appropriateness, feasibility), the mechanisms through which they may operate, and determinants (barriers and facilitators) of implementation that will inform future efforts to scale Bridges and other EE interventions.

Aim 4: Compare the cost and cost-effectiveness of the two implementation strategies. Using an activity-based ingredients approach, the investigators will examine how much each strategy costs to achieve a unit of effect.

ELIGIBILITY:
Inclusion Criteria:

Adolescent inclusion criteria:

1. Ages 11-17
2. a student at one of the 48 public primary schools included in the study-schools located in high HIV/AIDS prevalence areas in the greater Masaka region
3. living within a family and not an institution/orphanage

Caregiver inclusion criteria:

1. self-identified and confirmed by the adolescent and youth as primary caregiver of the adolescent and youth
2. capable of providing informed consent

Youth-serving NGOs inclusion criteria:

1. registered with the government of Uganda
2. willing to work with the study team
3. have a history of implementing micro-finance economic empowerment interventions.

Exclusion Criteria:

1. anyone with a significant cognitive impairment that interferes with their understanding of the informed consent process, or is unable/unwilling to consent.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1440 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Fidelity | Throughout intervention delivery (2 years (Baseline, 12 months, 24 months))
  The proportion of research assistants/facilitators that achieve 85% agreement on at least 3 of the fidelity assessment checklists.
  Field research assistants will be trained on using fidelity tools to track: (a) content of the intervention (e.g., saving), (b) process (e.g., mentoring skills), (c) activities (e.g., workshops). The team will practice fidelity assessment in pairs until they reach at least 85% agreement on at least 3 fidelity assessment checklists. In the field, independent fidelity observations will be conducted by research staff for 25% of Bridges sessions. Fidelity data will be used to assess the relationship between planned and actual implementation, and will be catalogued using FRAME-IS as a guide.
HIV prevalence | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Prevalence of adolescents positive for HIV among the sample determined from biomarker data

SECONDARY OUTCOMES:
Sexual risk-taking behavior | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Sexual risk-taking behavior will be measured using the Risk Behavior Survey. scores range from 0-20, with higher total scores indicating higher risk to engage in sexual risk behaviors.
Economic stability | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Economic stability will be assessed via Bank statements
School attainment | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  School attainment will be assessed using the Adapted Monitoring the Future scale and the Primary Leaving Examinations (PLE) Results
Depressive Symptoms | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Depressive symptoms was assessed using the Adapted Child Depression Inventory. The total score range between 0 and 28 with a high score indicating higher levels of depressive symptoms.
Proportion of adolescents living with HIV who are virally suppressed | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Viral suppression will be assessed using biological assay
Proportion of HIV negative adolescents who use PrEP | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  PrEP use will be assessed using biological assay
Hopelessness | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Hopelessness was assessed using the Beck Hopelessness Scale The total score range between 0 and 20 with a high score indicating higher levels of Hopelessness.
Self-Esteem | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Self-esteem was assessed using the Rosenberg Self-Esteems Scale. Scale scores range from 0 to 30 with higher scores indicative of higher self-esteem.
Self-concept | 4 years (Baseline, 12 months, 24 months, 36 months, 48 months post-baseline)
  Self-concept was assessed using the Tennessee Self-Concept Scale. Scale scores range from 20 to 100 with higher scores indicative of higher self-concept.

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Child Health and Development, Masaka, Uganda